CLINICAL TRIAL: NCT00917358
Title: Pegylated Interferon Alfa-2a for Dialysis Patients With Acute Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 940215
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Dialysis; Interferon
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pegylated interferon alfa-2a (Experimental): Pegylated interferon alfa-2a 135 ug/week for 24 weeks
  Interventions: Drug: Pegylated interferon alfa-2a
- Observation (No Intervention): Retrospectively chart review of dialysis patients with acute hepatitis C who did not receive any intervention

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a — Pegylated interferon alfa-2a 135 ug/week for 24 weeks
  Other Names: Pegylated interferon alfa-2a (Pegasys, Hoffman-La Roche)
  Arms: Pegylated interferon alfa-2a

SUMMARY:
Interferon-based monotherapy has been considered effective to treat acute hepatitis C in ordinary patients. However, the efficacy of this treatment has not been evaluated in prospective interventional studies for dialysis patients. The aim of the study is the evaluate the efficacy of peginterferon alfa-2a monotherapy for 24 weeks in this special clinical setting, and concomitantly evaluate retrospectively the dialysis patients with acute hepatitis C who did not receive intervention as the reference.

DETAILED DESCRIPTION:
Chronic viral hepatitis is common in dialysis patients, with the reported prevalence and annual incidence of 3-80% and 2.9%, respectively. The high incidence and prevalence in thse patients are attributed to potential nosocomial exposure to hepatitis C virus during dialysis, resulting in high rates of acute hepatitis C virus infection. It is estimated that about 65-80% of the patients who have acute hepatitis C will evolve to chronic infection, leading to chronic hepatitis, cirrhosis, hepatic decompensation, and hepatocellular carcinoma (HCC). Currently, interferon and pegylated interferon monotherapy remains effective to treat acute hepatitis C in ordinary patients, with the sustained virologic response (SVR) rates ranging from 65-90% after 12-24 weeks of therapy. However, few data regarding the efficacy and safety of interferon-based monotherapy is known till now. Treatment of weekly 135 pegylated interferon alfa-2a has shown superior safety to thrice weekly 3 million unit (MU) standard interferon alfa-2a for dialysis patients with chronic hepatitis C. Under the excellent safety profiles of treating dialysis patients with low dose pegylated interferon alfa-2a, we aimed to evaluate the efficacy of weekly 135 ug pegylated interferon alfa-2a for a total of 24 weeks for dialysis patients with acute hepatitis C, and also evaluate the SVR rate by retrospective chart review for dialysis patients with acute hepatitis C who did not receive interferon-based therapy to evaluate if early intervention for these patients will improve overall disease outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Creatinine clearance (Ccr) < 10 ml/min/1.73 m2
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive < 6 months with defined seroconversion
* Detectable serum quantitative HCV-RNA (Cobas Taqman HCV test, version 2, Roche Diagnostics) with a dynamic range of 25-391000000 IU/ml

Exclusion Criteria:

* Severe anemia (hemoglobin < 10 g/dL) or hemoglobinopathy
* Neutropenia (neutrophil count, <1,500/mm3)
* Thrombocytopenia (platelet <90,000/ mm3)
* Co-infection with HBV or HIV
* Chronic alcohol abuse (daily consumption > 20 g/day)
* Autoimmune liver disease
* Decompensated liver disease (Child classification B or C)
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception
* Unwilling to sign inform consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 1.0 year

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Chair — National Taiwan University Hospital; Jia-Horng Kao, MD, PhD, Principal Investigator — National Taiwan University Hospital; Cheng-Chao Liang, MD, Principal Investigator — Far Eastern Memorial Hospital; Shih-Jer Hsu, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch; Hung-Bin Tsai, MD, Principal Investigator — Buddhist Tzu Chi General Hospital; Peir-Haur Hung, MD, Principal Investigator — Chiayi Christian Hospital
Locations (5):
- Taiwan (5):
  - Buddhist Tzu Chi General Hospital, Chiayi City
  - Chiayi Christian Hospital, Chiayi City
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - National Taiwan University Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei